CLINICAL TRIAL: NCT00394147
Title: Phase II Trial of Pemetrexed and Gemcitabine in Patients With Advanced Head and Neck Cancer (SCCHN)
Brief Title: Pemetrexed and Gemcitabine in Patients With Advanced Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: stopped for lack of efficacy
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FER-HN-003
Record Dates: First submitted 2006-10-27; First posted 2006-10-31 (Estimated); Results first posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Head and Neck Cancer
Keywords: advanced; head; neck; cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasms | interventions — Pemetrexed; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pemetrexed and gemcitabine (Experimental): pemetrexed 500mg/m2 and gemcitabine 1500mg/m2 given on day 1 and day 15 of each 28 day cycle
  Interventions: Drug: pemetrexed; Drug: gemcitabine

INTERVENTIONS:
Drug: pemetrexed — pemetrexed 500mg/m2 given on day 1 and day 15 of each 28 day cycle
  Other Names: Alimta
Drug: gemcitabine — gemcitabine 1500mg/m2 given on day 1 and day 15 of each 28 day cycle
  Other Names: Gemzar

SUMMARY:
The purpose of this study is to look at how well the combination of two chemotherapy drugs, pemetrexed (Alimta) and gemcitabine (Gemzar) work to treat your cancer.

DETAILED DESCRIPTION:
This research study is being done because we have not yet been able to find the best treatment for recurrent or advanced head and neck cancer (SCCHN). Pemetrexed and gemcitabine have helped fight against SCCHN when each was given by itself. This study is different from others because it tests these two drugs together, which has not been tried before in patients with SCCHN. We will see how well these drugs can work to help to control or shrink your cancer.

We also want to find out what effects (good and bad) gemcitabine and pemetrexed have on you and your head and neck cancer. We do not know if these drugs will help you. Your cancer might get better or it might get worse. It might not have any effect on your condition. We can use what we learn from this research study to help other people with the same cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of squamous cell cancer of the head and neck - unresectable or metastatic. Must have measurable disease by RECIST.
* Karnofsky performance status greater than or equal to 60%
* Up to one prior systemic chemotherapy, immunotherapy allowed in the advanced or metastatic setting. This does not include prior chemotherapy, immunotherapy used with radiotherapy (ie concurrent with radiation therapy or as and induction regimen pror to definitive radiation therapy).
* At least 4 weeks from prior radiation or chemotherapy, must have recovered from all acute effects of treatment.
* Adequate organ and marrow function
* Negative pregnancy test. Agree to use birth control during and for 3 months after last dose of study drug.
* At least 18 years of age.
* Sign an informed consent and HIPAA consent.
* Must be able to take and absorb enteral medication.

Exclusion Criteria:

* Serious concomitant systemic disorder that would compromise safety or ability to complete study.
* Prior treatment with gemcitabine or pemetrexed within the previous year, unless used concurrently with radiation therapy.
* Pregnancy or breastfeeding.
* Symptomatic or uncontrolled brain mets. If treated, must be off steroids for at least 2 weeks.
* Inability or unwilling to take folic acid, vitamin B12, or dexamethasone.
* Treatment within last 30 days with a drug that has not received regulatory approval for any indication.
* Inability to interrupt and NSAID or salicylate with a long half-life (piroxicam or nabumetone) for a 5 day period.
* Presence of clinically relevant third space fluid that cannot be controlled by drainage or other procedure prior to study entry.
* Active, concurrent, invasive malignancy requiring ongoing treatment.
* Corticosteroids impermissible unless for adrenal failure, septic shock or as temporizing measure for symptomatic pain, breathing, or rash.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranee Mehra, MD, Principal Investigator — Fox Chase Cancer Center - Medical Oncology
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pemetrexed and Gemcitabine
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pemetrexed and Gemcitabine
Number analyzed (Participants) | 17
Age, Continuous [Median (Full Range); unit: years] | 64 [49 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pemetrexed and Gemcitabine
Number analyzed (Participants) | 17
Participants | 2

2. Secondary Outcome: Time to Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed and Gemcitabine
Number analyzed (Participants) | 17
months | 5.9 [.4 to 23.5]

3. Secondary Outcome: Overall Survival
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pemetrexed and Gemcitabine
Number analyzed (Participants) | 17
months | 5.9 [2.8 to 11.9]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Through study completion, an average of 1 year
Arm/Group | Pemetrexed and Gemcitabine
All-Cause Mortality (participants affected / at risk) | 14/17
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed and Gemcitabine (N=17)
Cellulitis (Infections and infestations) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Pain from worsening spinal metastases (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemetrexed and Gemcitabine (N=17)
Anemia (Blood and lymphatic system disorders) | 15
Pain (General disorders) | 12
Hyperglycemia (Metabolism and nutrition disorders) | 12
Fatigue (General disorders) | 11
Dysphagia (Gastrointestinal disorders) | 10
Cough (Gastrointestinal disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Nausea or vomiting (Gastrointestinal disorders) | 7
Xerostomia (Gastrointestinal disorders) | 7
Edema (General disorders) | 6
Insomnia (Psychiatric disorders) | 6
Myalgia arthralgia (Nervous system disorders) | 6
Dyspnea/Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 6
Alkaline phosphatase (Investigations) | 6
Increased LFTs (Investigations) | 6
Anorexia (Metabolism and nutrition disorders) | 6
White blood cell count decreased (Infections and infestations) | 5
Pruritis (Skin and subcutaneous tissue disorders) | 5
Fever (General disorders) | 4
Chills (General disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Dry cracked skin (Skin and subcutaneous tissue disorders) | 4
Heartburn (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Neuropathy- Sensory (Nervous system disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Mucositis (Gastrointestinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3
Hemorrhage (General disorders) | 3
Depression (Psychiatric disorders) | 3
Neuropathy-Motor (Nervous system disorders) | 3
Infection (w/o neutropenia) (Infections and infestations) | 3
Hypercalcemia (Investigations) | 3
Hyperkalemia (Investigations) | 3
Dysgeusia (Nervous system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 3
Orthostatic Hypotension (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Anxiety (Psychiatric disorders) | 2
Epiphora (Eye disorders) | 2
Weight Loss (Metabolism and nutrition disorders) | 2
Headache (Nervous system disorders) | 2
Creatinine (Renal and urinary disorders) | 2
Hypomagnesia (Investigations) | 2
Platelets (Blood and lymphatic system disorders) | 1
Dizziness (General disorders) | 1
Weakness (General disorders) | 1
Nail Changes (Skin and subcutaneous tissue disorders) | 1
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Infection with neutropenia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-01-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT00394147/Prot_SAP_000.pdf